CLINICAL TRIAL: NCT03932942
Title: Impact of Multiplex Respiratory Pathogen Testing on Antimicrobial Consumption and Hospital Admissions at Pediatric Emergency Room: A Randomized Controlled Trial
Brief Title: Point-of-care Testing of Respiratory Pathogens at Pediatric Emergency Room
Acronym: Hevi-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EETTMK_08_2019
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Tract Infections
Keywords: Anti-bacterial agents; Emergency room; Respiratory pathogen; Point-of-care testing; Patient admission; Pediatrics; Pediatric emergency medicine; Cost-benefit analysis; Antimicrobial stewardship
MeSH Terms: conditions — Respiratory Tract Infections; Emergencies

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial 2:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care testing of respiratory pathogens on admission (Experimental): Point-of-care testing of respiratory pathogens on admission. The subjects will receive the point-of-care testing of respiratory pathogens at pediatric emergency room. The results are ready within 1 one hour.
  Interventions: Diagnostic Test: QIAstat at pediatric emergency room
- Routine ED protocol (No Intervention): Diagnostic tests for respiratory pathogens will be obtained according to clinical judgement and tested on microbiological laboratory. The results are ready on the next office day.

INTERVENTIONS:
Diagnostic Test: QIAstat at pediatric emergency room — Pediatric acute care nurses will obtain respiratory samples for testing from all patients with fever or any respiratory symptom.
  Arms: Point-of-care testing of respiratory pathogens on admission

SUMMARY:
The main objective of the trial is to evaluate the effect of point-of-care testing of respiratory pathogens at a pediatric emergency room on the antibiotic consumption and hospital admissions in acutely ill children.

DETAILED DESCRIPTION:
The study is a randomized controlled trial including children 0 up to 17 years of age with fever or acute respiratory infection at a pediatric emergency department in university hospital. In total 1668 subjects will be randomly allocated to undergo point-of-care multiplex respiratory pathogen testing with results ready within approximately one hour or to a control group with testing according to clinical judgement and results ready within next office day. Subjects will be randomized on admission and unequal allocation ratio of 2:1 (1112 subjects to intervention and 556 subjects to control arm) will be used. Data on rate of hospitalization, antibiotic prescriptions, ancillary testing and length of visit will be collected using medical record system.

ELIGIBILITY:
Inclusion Criteria:

* Any respiratory symptom defined as tachypnea, shortness of breath, apnea, wheezing, cough, rhinitis, croup, sneezing, ear ache, or sore throat AND/OR
* Fever > 38.0 C

Exclusion Criteria:

* Need of resuscitation at emergency room
* Need of immediate transfer to pediatric intensive care unit

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1350 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Proportion of children with antibiotic prescription at emergency room | Up to 1 day after study entry
  Antibiotic consumption at emergency room

SECONDARY OUTCOMES:
Proportion of children with antibiotics in one week | 0-7 days after study entry
  Antimicrobial prescription rate
Proportion of children receiving macrolide antibiotic at pediatric emergency room | Up to 1 day after study entry
  Among all children randomized
Proportion of infants aged < 3 months receiving macrolide antibiotic at pediatric emergency room | Up to 1 day after study entry
  Among all children randomized
Proportion of children admitted to hospital | Up to 1 day after study entry
  Hospital admissions
Proportion of children admitted to hospital | 0-7 days after study entry
  Hospital admissions
Number of other diagnostic tests than point-of-care test performed at emergency room | Up to 1 day after study entry
  Number and cost of diagnostic tests such as blood culture, blood chemistry
Proportion of children with readmission to hospital or revisit at emergency room | 0-7 days after study entry
  Proportion of children with hospital readmission or emergency room revisit within 7 days after discharge from ED or hospital
Proportion of children with outpatient telephone contact within 7 days after discharge from emergency room | 0-7 days
  Outpatient telephone contact within 7 days after discharge from emergency room
Number of diagnostic tests per child other than point-of-care test performed within one week | 0-7 days after discharge
  Ancillary laboratory testing
Proportion of children with admission to pediatric intensive care unit or intensive care unit | 0-30 days
  Admission to pediatric intensive care unit or intensive care unit
Proportion of children who died within one month after study entry | 0-30 days
  Mortality
Cost in euros per child per visits | 0-7 days after study entry
  Visit associated cost (euros)
Length of stay at emergency room in minutes | Up to 1 day after study entry
  Mean length of visit at emergency room (minutes)
Proportion of children receiving correct pathogen directed therapy | 0-7 days after study entry
  Antimicrobial use for Mycoplasma pneumoniae, pertussis and influenza
Time to initiation of correct pathogen directed therapy | 0-7 days after study entry
  Antimicrobials for Mycoplasma pneumoniae, pertussis and influenza (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Terhi S Tapiainen, MD,PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Department of Pediatrics, Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared according to the practice in place at the time of the study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the study completion or at submission
Access Criteria: For reviewers and editors before publishing and after publishing for the whole research community

REFERENCES:
- [Derived] Mattila S, Paalanne N, Honkila M, Pokka T, Tapiainen T. Effect of Point-of-Care Testing for Respiratory Pathogens on Antibiotic Use in Children: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2216162. doi: 10.1001/jamanetworkopen.2022.16162. PMID 35679047